CLINICAL TRIAL: NCT05719584
Title: Effects of Pelvic Floor Muscle Training With and Without Hypopressive Exercises on Pelvic Organ Prolapse in Postmenopausal Females.
Brief Title: Pelvic Floor Muscle Training With and Without Hypopressive Exercises in Postmenopausal Females.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0502
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Pelvic Organ Prolapse
Keywords: pelvic organ prolapse; postmenopausal; females; exercises
MeSH Terms: conditions — Pelvic Organ Prolapse; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hypopressive exercises (Experimental): pelvic floor muscle exercises along with hypopressive exercises
  Interventions: Other: hypopressive exercises; Other: pelvic floor muscle training
- pelvic floor muscle training (Active Comparator): pelvic floor muscle exercises alone
  Interventions: Other: pelvic floor muscle training

INTERVENTIONS:
Other: hypopressive exercises — patients will receive pelvic floor muscle training with hypopressive exercises at outpatient department. Treatment will continue for 12 weeks 3 days per week. They will receive information about the localization and function of the PFM and transversus abdominis (TrA) muscles. Next, lying in a supine position with flexed knees and hips, they will localize their own pelvic floor with the help of touching their perineum. Then they will be instructed how to contract the PFM correctly, then they will directed to contract PFMs and in the end participants will be taught how to voluntarily contract the PFM simultaneously with diaphragmatic Aspiration(8-10 repetitions daily
  Arms: hypopressive exercises
Other: pelvic floor muscle training — patients will receive only pelvic floor muscle training exercises(pelvic floor muscle contractions) at the outpatient department and treatment will continue for 12 weeks 3 days per week. PFMT will be performed in the lying, sitting and standing positions. The patients will be instructed to perform three sets of 8-12 maximum voluntary contractions held for 6 sec, with 12 sec of rest between each contraction, followed by three fast contractions in a row

SUMMARY:
To compare the effects of pelvic floor muscle training with and without hypopressive exercises on pelvic organ prolapse in postmenopausal females

DETAILED DESCRIPTION:
In this randomized controlled trial multigravida, postmenopausal females with stage 1 and 2 pelvic organ prolapse will be taken (exclusion criteria includes cesarean section females, ovarian cysts ,UTIs and neoplasm). This study will be conducted in Jinnah hospital , Lahore. Sample size of 36 will be taken according to inclusion criteria. Study will be completed in 10 months after approval of synopsis. Non-Probability convenient sampling will be used. A written consent form will be taken from participants meeting inclusion criteria and will be randomly allocated into two groups through lottery method, to either the Pelvic floor muscle training group or group with combined pelvic floor muscle exercise and hypopressive exercise. Treatment period will be 12 weeks 3 days per week. The participants will be advised not to use other forms of treatment during the trial (pharmacologic or non pharmacologic treatment). All subjects will be assessed before and after treatment by POP-Q, pelvic floor impact questionnaire and P-QOL. Data will be analyzed by using SPSS 25 statistical software.

ELIGIBILITY:
Inclusion Criteria:

* Multigravida
* Previous spontaneous vaginal deliveries
* Diagnosed Stage 1 and 2 pelvic organ prolapse
* Post-menopausal females

Exclusion Criteria:

* History of cesarean section
* History of ovarian cysts
* History of UTIs
* History of neoplasm
* Instrumental deliveries

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — postmenopausal females
Enrollment: 36 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
pelvic organ prolapse quantification (POP-Q) | 12th week
  POP-Q can be seen in Many clinical settings & published researches and it is used to grade and measure of pelvic organ prolapse during its assessment.
Pelvic Floor Impact Questionnaire-7 (PFIQ-7) | 12th week
  It is a short and less comprehensive version of Pelvic Floor Impact Questionnaire (PFIQ). It is a health related questionnaire for women with pelvic floor conditions.
  consists of 7 questions that need to be answered 3 times each.
Prolapse Quality of life questionnaire(P-QOL) | 12th week
  A simple, valid, reliable questionnaire to assess the severity of symptoms and their impact on the quality of life in women with Pelvic organ prolapse. There are several questions which a participant needs to answer.

CONTACTS AND LOCATIONS:
Overall Officials: hina gul, MS-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Jinnah hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nam G, Lee SR, Choi S. Clitoromegaly, Vulvovaginal Hemangioma Mimicking Pelvic Organ Prolapse, and Heavy Menstrual Bleeding: Gynecologic Manifestations of Klippel-Trenaunay Syndrome. Medicina (Kaunas). 2021 Apr 9;57(4):366. doi: 10.3390/medicina57040366. PMID 33918633
- [Background] Alves FK, Riccetto C, Adami DB, Marques J, Pereira LC, Palma P, Botelho S. A pelvic floor muscle training program in postmenopausal women: A randomized controlled trial. Maturitas. 2015 Jun;81(2):300-5. doi: 10.1016/j.maturitas.2015.03.006. Epub 2015 Mar 14. PMID 25862491
- [Background] Barber MD. Pelvic organ prolapse. BMJ. 2016 Jul 20;354:i3853. doi: 10.1136/bmj.i3853. No abstract available. PMID 27439423
- [Background] Fatima Q, Razzaqe H, Kashif M, Aslam F. Association of parity and pelvic organ prolapse. Journal of Rawalpindi Medical College Students Supplement. 2016;20:104-8.
- [Background] Resende APM, Bernardes BT, Stupp L, Oliveira E, Castro RA, Girao MJBC, Sartori MGF. Pelvic floor muscle training is better than hypopressive exercises in pelvic organ prolapse treatment: An assessor-blinded randomized controlled trial. Neurourol Urodyn. 2019 Jan;38(1):171-179. doi: 10.1002/nau.23819. Epub 2018 Oct 12. PMID 30311680
- [Background] Parle J, Shahmalak S, Irkar D. Effect of Hypopressive exercise in women with Pelvic Organ Prolapse. Nepal Journal of Obstetrics and Gynaecology. 2021;16(1).
- [Background] Fleischer K, Thiagamoorthy G. Pelvic organ prolapse management. Post Reprod Health. 2020 Jun;26(2):79-85. doi: 10.1177/2053369120937594. PMID 32627701
- [Background] Navarro-Brazalez B, Prieto-Gomez V, Prieto-Merino D, Sanchez-Sanchez B, McLean L, Torres-Lacomba M. Effectiveness of Hypopressive Exercises in Women with Pelvic Floor Dysfunction: A Randomised Controlled Trial. J Clin Med. 2020 Apr 17;9(4):1149. doi: 10.3390/jcm9041149. PMID 32316686
- [Background] Navarro Brazalez B, Sanchez Sanchez B, Prieto Gomez V, De La Villa Polo P, McLean L, Torres Lacomba M. Pelvic floor and abdominal muscle responses during hypopressive exercises in women with pelvic floor dysfunction. Neurourol Urodyn. 2020 Feb;39(2):793-803. doi: 10.1002/nau.24284. Epub 2020 Jan 27. PMID 31985114
- [Background] Juez L, Nunez-Cordoba JM, Couso N, Auba M, Alcazar JL, Minguez JA. Hypopressive technique versus pelvic floor muscle training for postpartum pelvic floor rehabilitation: A prospective cohort study. Neurourol Urodyn. 2019 Sep;38(7):1924-1931. doi: 10.1002/nau.24094. Epub 2019 Jul 11. PMID 31297874
- See also: A study conducted in 2023 by Guadalupe Molina-Torres et al, was to assess the effects of an 8-week, highly supervised programme of hypopressive exercises on the strength of the pelvic floor muscles and the signs and symptoms of urinary incontinence. — https://pubmed.ncbi.nlm.nih.gov/36482844/